CLINICAL TRIAL: NCT01324024
Title: Attention & Memory Impairments in Menopausal Women: A Possible Role for Vyvanse?
Brief Title: Attention & Memory Impairments in Menopausal Women
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Shire (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 812470
Record Dates: First submitted 2011-03-24; First posted 2011-03-28 (Estimated); Results first posted 2017-06-28 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-05

CONDITIONS: Symptomatic Menopause; Cognitive Impairments
Keywords: Menopause; Aging; Memory; Women
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Lisdexamfetamine Dimesylate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lisdexamfetamine, then placebo (Experimental): Participants first received titrated doses of Lisdexamfetamine 20 to 60 mg/d each day for 4 weeks followed by a 2-week washout, then they received Placebo tablets (matching Lisdexamfetamine tablets) each day for 4 weeks.
  Interventions: Drug: Lisdexamfetamine; Drug: Placebo
- Placebo, then Lisdexamfetamine (Experimental): Participants first received Placebo tablets (matching Lisdexamfetamine tablets) each day for 4 weeks followed by a 2-week washout, then they received titrated doses of Lisdexamfetamine 20 to 60 mg/d each day for 4 weeks.
  Interventions: Drug: Lisdexamfetamine; Drug: Placebo

INTERVENTIONS:
Drug: Lisdexamfetamine — In a counterbalanced fashion, participants would receive titrated doses of LDX 20 to 60 mg/d for 4 weeks followed by a 2-week washout and then crossed over to the placebo tablets for another 4 weeks. All women will start with LDX 20 mg/d and then be titrated to 40 mg/d after 1 week and 60 mg/d after 2 weeks (as tolerated).
  Other Names: Vyvanse®
Drug: Placebo — In a counterbalanced fashion, participants would receive placebo tablets for 4 weeks followed by a 2 week washout, then will receive titrated doses of LDX 20 to 60 mg/d for 4 weeks.

SUMMARY:
The purpose of this study is to determine whether a medication called Vyvanse® (lisdexamfetamine; LDX) has an impact on cognitive functioning, specifically measures of sustained attention, verbal encoding and recall and working memory, in menopausal aged women. LDX is a medication used to treat attention deficit hyperactivity disorder (ADHD). The cognitive difficulties that menopausal women report experiencing are typical of adults who are diagnosed with ADHD. The investigators will assess whether or not LDX is effective in alleviating those cognitive disruptions when compared to a placebo.

DETAILED DESCRIPTION:
Midlife decline in cognitive function, particularly attention and working memory, is a frequent complaint for which menopausal women seek clinical intervention. Many of the cognitive complaints detected in menopausal women including, short-term memory, organization of tasks, sustaining focus and concentration, and regulating emotions, overlap with symptoms frequently reported by adults with ADHD. These impairments are reported by many women who have no previous history of ADHD, and appear to be linked to reduced estrogen levels occurring in menopause.

This is a double-blind, placebo-controlled, cross-over study testing whether LDX, a stimulant medication, would be effective in alleviating midlife onset impairments of attention and working memory among menopausal women. There will be 3 days in which subjects will undergo a brief cognitive testing assessment; the first testing period will occur at baseline prior to beginning LDX or placebo treatment (PT) in trial A; the second testing period will occur following 4 weeks of double blind LDX or PT; and the final testing period will take place after another 4 weeks of double blind LDX or PT in Trial B. Each cognitive test period will involve 2 separate cognitive testing batteries that will take approximately 120 minutes total to complete.

ELIGIBILITY:
Inclusion Criteria:

Women ages 45 to 60 will be eligible for this study if they:

* Are within 5 years of their last menstrual period;
* Are able to give written informed consent;
* Must have clear urine toxicology screen upon recruitment;
* Are fluent in written and spoken English;
* Must have negative urine pregnancy test if still menstruating.

Exclusion Criteria:

* History of seizures;
* History of cardiac disease including known cardiac defect or conduction abnormality;
* Abnormal electrocardiogram during screening;
* Use of estrogen therapy within previous 6 months;
* Current pregnancy or planning to become pregnant.
* Presence of a contraindication to treatment with stimulant medication; this would include the presence of hypertension, coronary disease, atrial fibrillation, and arrhythmia.

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2011-05; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia N Epperson, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- Penn Center for Women's Behavioral Wellness, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Epperson CN, Pittman B, Czarkowski KA, Bradley J, Quinlan DM, Brown TE. Impact of atomoxetine on subjective attention and memory difficulties in perimenopausal and postmenopausal women. Menopause. 2011 May;18(5):542-8. doi: 10.1097/gme.0b013e3181fcafd6. PMID 21293309
- [Result] Epperson CN, Shanmugan S, Kim DR, Mathews S, Czarkowski KA, Bradley J, Appleby DH, Iannelli C, Sammel MD, Brown TE. New onset executive function difficulties at menopause: a possible role for lisdexamfetamine. Psychopharmacology (Berl). 2015 Aug;232(16):3091-100. doi: 10.1007/s00213-015-3953-7. Epub 2015 Jun 11. PMID 26063677
- See also: Click here for more information about our center. — http://www.med.upenn.edu/womenswellness/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 55 participants were consented for screening over the course of 2 years at an outpatient research site in Philadelphia, PA.
Pre-assignment Details: Of the 55 who were consented for screening, 20 did not meet inclusion criteria and of the remaining 35, 32 participants completed the study.
Groups:
- Lisdexamfetamine, Then Placebo: Participants first received titrated doses of Lisdexamfetamine 20 to 60 mg/d each day for 4 weeks (i.e, 20mg/d for 1 week, 40mg/d for 1 week and 60mg/d for 2 weeks) followed by a 2-week washout, then they received Placebo tablets (matching Lisdexamfetamine tablets) each day for 4 weeks.
- Placebo First, Then Lisdexamfetamine: Participants first received Placebo tablets (matching Lisdexamfetamine tablets) each day for 4 weeks, followed by a 2-week washout, then they received titrated doses of Lisdexamfetamine 20 to 60 mg/d each day for 4 weeks (i.e, 20mg/d for 1 week, 40mg/d for 1 week and 60mg/d for 2 weeks).
Period: First Intervention (4 Weeks)
Arm/Group | Lisdexamfetamine, Then Placebo | Placebo First, Then Lisdexamfetamine
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0
Period: Washout (2 Weeks)
Arm/Group | Lisdexamfetamine, Then Placebo | Placebo First, Then Lisdexamfetamine
Started | 18 | 17
Completed | 18 | 17
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Lisdexamfetamine, Then Placebo | Placebo First, Then Lisdexamfetamine
Started | 18 | 17
Completed | 16 | 16
Not Completed | 2 | 1
Not completed — Withdrawal by Subject | 2 | 1

BASELINE CHARACTERISTICS:
Population: Of the 55 subjects who were consented for screening, 20 were excluded and of the remaining 35 subjects, 32 completed both active and placebo treatment trials. There were 3 subjects who withdrew themselves from the study. These 3 subjects are not included in the overall number of baseline participants analyzed.
Groups:
- All Study Participants: Participants were randomized to receive either Lisdexampethamine in titrated doses (20mg/d- 60mg/d) or Placebo tablets (matching Lisdexamphetamine).
Arm/Group | All Study Participants
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 22
  More than one race | 2
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 32

OUTCOME MEASURES:

1. Primary Outcome: Brown Attention Deficit Disorder Scale (BADDS)
Description: The BADDS questionnaire is a clinician administered questionnaire that assesses the frequency and severity of five clusters of symptoms reflective of executive dysfunction reported by individuals with ADHD. Participants are asked to rate the frequency and severity of a symptom on a scale from 0 to 3, with 0 meaning that the problem described does not relate to them and 3 indicating that the problem is very true for them and occurs almost daily. The range of severity for the total BADDS score is 0 to 120, with scores of 55 and above being consistent with full-syndrome ADHD.
Time Frame: Baseline, end of first Intervention (4 weeks) and end of second Intervention (4 weeks)
Population: Of the 55 participants who were consented for screening, 20 were excluded. Of the remaining 35 subjects, 32 completed both active and placebo treatment trials. The numbers in the lisdexamphetamine and placebo arms reflect the fact that 32 subjects completed both arms. 35 total participant data was analyzed for the baseline arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lisdexamfetamine: Participants who received Lisdexamfetamine 20
- Sugar Pill: Placebo pill, capsules
  Lisdexamfetamine: The purpose of this study is to assess whether or not lisdexamfetamine is effective in alleviating cognitive disruptions when compared to a placebo.
Arm/Group | Baseline | Lisdexamfetamine | Sugar Pill
Number analyzed (Participants) | 35 | 32 | 32
units on a scale | 35.7 (16.8) | 21.2 (16.8) | 29.8 (17.7)

2. Secondary Outcome: Penn Continuous Performance Test
Description: The Penn Continuous Performance Test is a measure of visual attention and vigilance. In this task, a series of red vertical and horizontal lines flash in a digital numeric frame. The participant must press the spacebar whenever the lines form complete numbers or complete letters. The minimum to maximum score range for this task is 0-60 correct responses, with 60 being a perfect score. This data presented in the outcome measure table reflects the total number of correct responses.
Time Frame: Baseline, end of first Intervention (4 weeks) and end of second Intervention (4 weeks)
Population: The numbers in the lisdexamphetamine and placebo arms reflect the fact that 32 subjects completed both arms; 16 participants in each arm. 35 total participant data was analyzed for the baseline arm.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lisdexamfetamine: Lisdexamfetamine or Vyvanse
  Lisdexamfetamine: The purpose of this study is to assess whether or not lisdexamfetamine is effective in alleviating cognitive disruptions when compared to a placebo.
Arm/Group | Baseline | Lisdexamfetamine | Sugar Pill
Number analyzed (Participants) | 35 | 32 | 32
units on a scale | 53.29 (3.78) | 56.37 (3.59) | 56.21 (3.27)

3. Secondary Outcome: NYU Paragraph Recall Task
Description: Subjects hear 2 brief narratives, each containing 19-21 informational bits, and are asked to recall as many details as possible immediately after hearing each paragraph (A and B) and again following a 30 minute delay. Subjects receive credit for each informational bit recalled verbatim. Different paragraphs were read at each assessment. The maximum number of correct responses for paragraph A is 19 and the maximum number of correct responses for paragraph B is 21.
Time Frame: Baseline, end of first Intervention (4 weeks) and end of second Intervention (4 weeks)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Lisdexamfetamine: Participants received titrated doses of Lisdexamfetamine 20 to 60 mg/d each day for 4 weeks (i.e, 20mg/d for 1 week, 40mg/d for 1 week and 60mg/d for 2 weeks).
- Placebo: Participants received Placebo tablets (matching Lisdexamfetamine tablets) each day for 4 weeks.
Arm/Group | Baseline | Lisdexamfetamine | Placebo
Number analyzed (Participants) | 35 | 32 | 32
units on a scale
  Immediate paragraph recall A | 7.09 (2.56) | 7.48 (2.63) | 7.00 (2.70)
  Immediate paragraph recall B | 6.38 (2.12) | 7.45 (3.20) | 6.75 (2.53)
  Delayed paragraph recall A | 4.68 (2.65) | 5.90 (3.38) | 4.94 (3.02)
  Delayed paragraph recall B | 7.81 (3.58) | 9.77 (3.53) | 8.47 (2.97)

ADVERSE EVENTS:
Time Frame: From study start to study completion only
Arm/Group | Lisdexamfetamine | Sugar Pill
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 6/32 | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lisdexamfetamine (N=32) | Sugar Pill (N=32)
diverticulitis (Gastrointestinal disorders) | 2 (2) | 0 (0) — 2 participants experienced symptoms of diverticulitis while on active study drug. Both were hospitalized for a day or less. One received antibiotic treatment and both stopped drug for a short period of time.
increased heart rate (Cardiac disorders) | 1 (1) | 1 (1) — One subject experienced an increased heart in response to the active study drug.
mouth sensitivity (General disorders) | 2 (2) | 0 (0) — 2 subjects experienced gum and tongue sensitivity while on active study drug.
dizziness (General disorders) | 0 (0) | 1 (1) — One subject experienced dizziness in response to placebo pill.
eye irritation (Eye disorders) | 1 (1) | 0 (0) — One subject experienced eye irritation in response to active study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes